CLINICAL TRIAL: NCT05990231
Title: Cadonilimab Combined With Anlotinib in Locally Advanced or Relapsed/Metastatic Esophageal Squamous Cell Carcinoma Patients After Failure of PD-1 Inhibitor Combined With Platinum-containing Chemotherapy: A Single-center, Single-arm Exploratory Study
Brief Title: Cadonilimab/Anlotinib in Locally Advanced or Relapsed/Metastatic ESCC Patients After Failure of PD-1 Combined With Platinum-containing Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0563
Record Dates: First submitted 2023-08-06; First posted 2023-08-14 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-08

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Esophageal Squamous Cell Carcinoma; Cadonilimab; Anlotinib; CTLA-4; PD-1
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Diabetes Mellitus, Insulin-Dependent, 12

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cadonilimab combined with anlotinib (Experimental)
  Interventions: Drug: Cadonilimab combined Anlotinib

INTERVENTIONS:
Drug: Cadonilimab combined Anlotinib — Cadonilimab: intravenous administration at a dose of 10mg/kg on day 1 of each cycle, every 3 weeks (Q3W) Anlotinib: 12mg, orally once a day (orally before breakfast, the daily medication time should be as the same as possible), continuous taking for 2 weeks, stopping for 1 week, 3 weeks (21 days) as a treatment cycle

SUMMARY:
Advanced esophageal squamous cell carcinoma patients who have failed first-line PD-1 inhibitor combined with chemotherapy lack a standard treatment option. Second-line treatments have limited efficacy, indicating a significant unmet clinical need. Anlotinib is a novel multi-target tyrosine kinase inhibitor (TKI) has anti-tumor angiogenesis and tumor growth inhibition effects. Cadonilimab is a human immunoglobulin (Ig) G1 monoclonal antibody (mAb), which is a bispecific antibody that blocks both PD-1 and CTLA-4. Both of them have shown certain efficacy and good safety in more than second-line therapy for patients with advanced esophageal squamous cell carcinoma as monotherapy. This study aims to evaluate the efficacy and safety of cadonilimab combined with anlotinib in patients with locally advanced or recurrent/metastatic esophageal squamous cell carcinoma who have progressed on PD-1 inhibitor combined with platinum-containing chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign a written informed consent form.
2. Age ≥18 and ≤80 years, both males and females are eligible.
3. ECOG performance status score of 0 or 1.
4. Expected survival≥3 months.
5. Patients with locally advanced or recurrent/metastatic esophageal squamous cell carcinoma confirmed by histology and/or cytology that is incurable (including curative surgery and curative radio/chemotherapy). Patients with locally advanced or recurrent/metastatic esophageal squamous cell carcinoma who have failed of PD-1 inhibitor combined with platinum-based chemotherapy , and are not allowed to receive other systemic anti-tumor treatments. Note: For patients who have received adjuvant/neoadjuvant PD-1 inhibitor combined with platinum-based chemotherapy for non-metastatic disease with curative intent, or curative platinum-based radio/chemotherapy combined with PD-1 inhibitor for locally advanced or recurrent/metastatic disease, if disease progression occurs within <6 months after the end of the last treatment, and the patients has not received other systemic anti-tumor treatments after disease progression, they are allowed to be enrolled.
6. According to RECIST v1.1, patients must have at least one measurable lesion. For patients who have received radiotherapy previously and have no other target lesions available, when there is objective evidence of significant progression after radiotherapy, the lesion treated with radiotherapy can be considered as a target lesion.
7. The function of important organs meets the following requirements (excluding any blood components and growth factors used within 14 days):

   1. Normal bone marrow function, neutrophils ≥1,500/mm3, platelet count ≥100,000/mm3, hemoglobin ≥5.6 mmol/L (9g/dL);
   2. Normal renal function or serum creatinine ≤1.5 mg/dL and/or creatinine clearance rate ≥60 ml/min;
   3. Normal liver function or bilirubin ≤1.5 times ULN, ASAT & ALST ≤1.5 times ULN.
8. Female patients of childbearing potential must undergo a urine or serum pregnancy test within the first 3 days before the first dose (if the urine pregnancy test result cannot be confirmed as negative, a serum pregnancy test must be performed, and the serum pregnancy result will prevail), and the result must be negative. If a female patient of childbearing potential has sexual intercourse with an uncircumcised male partner, the subject must take effective contraceptive measures from the beginning of screening and must agree to continue using contraceptive methods for 120 days after the last dose of study drug; whether to stop contraception after this time point should be discussed with the investigator.
9. If an uncircumcised male subject has sexual intercourse with a female partner of childbearing potential, the subject must take effective contraceptive measures from the beginning of screening until 120 days after the last dose; whether to stop contraception after this time point should be discussed with the investigator.
10. The patient is willing and able to comply with the scheduled visits, treatment plan, laboratory tests, and other requirements of the study.

Exclusion Criteria:

Subjects who meet any of the following criteria will be ineligible to participate in this study:

1. Subjects who have had other malignant tumors within 3 years prior to enrollment, except those who have been cured by local treatment such as basal or squamous cell skin cancer, superficial bladder cancer, cervical or breast carcinoma in situ.
2. Subjects who are concurrently enrolled in another clinical study, unless it is an observational, non-interventional clinical study or a follow-up period of an interventional study.
3. Subjects who have received systemic anti-tumor therapy (chemotherapy, immunotherapy, etc.) for non-target lesions within 3 weeks before the first dose of study drug; palliative local therapy for non-target lesions within 2 weeks before the first dose of study drug; non-specific immunomodulatory therapy (such as interleukin, interferon, thymosin, tumor necrosis factor, etc., excluding IL-11 for thrombocytopenia) within 2 weeks before the first dose of study drug; or Chinese herbal medicine or traditional Chinese medicine with anti-tumor indications within 1 week before the first dose of study drug.
4. Subjects who have received any treatment targeting tumor immune mechanisms, such as immunotherapy other than PD-1 inhibitors (including immune checkpoint inhibitors such as anti-CTLA-4 antibodies, anti-CD47 antibodies, anti-SIRPα antibodies, anti-LAG-3 antibodies, etc.), immune checkpoint agonists (such as ICOS, CD40, CD137, GITR, OX40 antibodies, etc.), immune cell therapy, biologics, etc., other than PD-1 inhibitors.
5. Subjects who have experienced any of the following during previous PD-1 inhibitor treatment:

   1. Grade 3 or higher irAE caused by PD-1 inhibitor treatment (excluding endocrine system-related irAEs), irAEs that led to permanent discontinuation of treatment, grade 2 immune-related cardiac toxicity or any grade of neurologic or ophthalmologic irAE.
   2. All adverse events during previous PD-1 inhibitor treatment have not been completely resolved or resolved to grade 1 before screening for this study. For subjects with grade ≥2 endocrine adverse events, if the condition is stable with appropriate alternative treatment and asymptomatic, enrollment is allowed.
   3. Previous adverse events that required the use of immunosuppressive agents other than glucocorticoids or recurrence of adverse events during previous immunotherapy that required systemic use of glucocorticoids.
6. Screening imaging shows that the tumor surrounds or invades important blood vessels or organs (such as the heart and pericardium, trachea, aorta, superior vena cava, etc.), or there is obvious necrosis or cavity, and the investigator judges that entering the study would increase the risk of bleeding; there are subjects at risk of developing esophagotracheal fistula or esophageal pleural fistula.
7. Subjects who have had active autoimmune diseases requiring systemic treatment in the past two years (such as use of disease-modifying drugs, corticosteroids, immunosuppressive therapy), and replacement therapy (such as thyroid hormone, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered systemic treatment.
8. Subjects with non-infectious pneumonia/interstitial lung disease (including radiation pneumonitis) requiring systemic glucocorticoid therapy that is currently uncontrolled.
9. Presence of brainstem, meningeal metastasis, spinal cord metastasis or compression.
10. Presence of active central nervous system (CNS) metastatic lesions. Note: Subjects with previously treated brain metastases (such as surgery or radiotherapy) are allowed to enroll if they are clinically stable for at least 2 weeks (from the time of first administration of study drug) and have discontinued corticosteroid hormones for 7 days before administration of study drug; untreated asymptomatic brain metastases (i.e., no neurological symptoms, no need for corticosteroid hormones, no brain metastases with a long axis >1.5 cm and no obvious peritumoral edema) are eligible to enroll.
11. Presence of pleural effusion, pericardial effusion or ascites with clinical symptoms or requiring repeated drainage.
12. Presence of uncontrolled comorbidities currently including but not limited to decompensated liver cirrhosis, nephrotic syndrome, uncontrolled metabolic disorders, or psychiatric/social conditions that would limit compliance with study requirements or affect the subject's ability to provide written informed consent.
13. History of myocarditis, cardiomyopathy or malignant arrhythmia. Unstable angina pectoris requiring hospitalization within 12 months before the first dose of study drug, myocardial infarction, congestive heart failure (New York Heart Association functional class II or higher), vascular disease (such as aortic aneurysm at risk of rupture), or other cardiac damage that may affect the safety evaluation of the study drug (such as poorly controlled arrhythmia or myocardial ischemia) within 12 months before the first dose of study drug.
14. Occurrence of any arterial thrombotic events within 6 months before the first dose of study drug; grade 3 or higher venous thromboembolic events according to NCI CTCAE 5.0; transient ischemic attacks; cerebrovascular accidents; hypertensive crises or hypertensive encephalopathy; exacerbation of chronic obstructive pulmonary disease within 1 month before the first dose of study drug; current hypertension with systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg despite oral antihypertensive therapy.
15. History of severe bleeding tendency or coagulation dysfunction; significant bleeding symptoms within 1 month before the first dose of study drug, including but not limited to gastrointestinal bleeding, bleeding peptic ulcer, hemoptysis (defined as coughing up or spitting out ≥1 teaspoon fresh blood or small clots or coughing up blood without sputum), which allows for inclusion if it is due to hemorrhoids and does not require intervention.
16. Active or past history of confirmed inflammatory bowel disease (such as Crohn's disease, ulcerative colitis, or chronic diarrhea).
17. Severe infection occurring within 4 weeks prior to the first dose of study drug, including but not limited to complications requiring hospitalization, sepsis, or severe pneumonia; active infection treated with systemic anti-infective therapy within 2 weeks prior to the first dose of study drug (excluding antiviral therapy for hepatitis B or C).
18. Known active tuberculosis (TB) or suspected active TB requiring clinical evaluation to rule out; known active syphilis infection.
19. Participants with active hepatitis B (HBsAg-positive with HBV-DNA levels above 1000 copies/mL (200 IU/mL) or higher than the lower limit of detection, whichever is higher) must receive antiviral therapy for hepatitis B during the study treatment period; active hepatitis C infection (HCV antibody-positive with HCV-RNA levels above the lower limit of detection).
20. History of immunodeficiency; positive HIV antibody test; current use of long-term systemic corticosteroids or other immunosuppressive agents.
21. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
22. Unresolved toxicities from prior anti-tumor therapy, defined as toxicities not yet resolved to NCI CTCAE version 5.0 grade 0 or 1, or at a level dictated in the inclusion/exclusion criteria, with the exception of alopecia. Participants with irreversible toxicities that are not expected to be exacerbated by study drug may be included in the study after consultation with the investigator (e.g., hearing loss). Participants with radiation-induced long-term toxicities judged by the investigator to be irreversible may be included in the study.
23. Major surgery or serious injury within 30 days prior to the first dose of study drug, or planned major surgical procedure within 30 days after the first dose of study drug (at the discretion of the investigator); minor surgical procedure within 3 days prior to the first dose of study drug (excluding peripheral venous catheterization and placement of venous infusion port).
24. Known hypersensitivity to any component of the study drug; history of serious hypersensitivity reaction to other monoclonal antibodies.
25. Receipt of live vaccine or attenuated live vaccine within 30 days prior to the first dose of study drug, or planned receipt of live vaccine or attenuated live vaccine during the study period; use of inactivated vaccine is allowed.
26. Known history of psychiatric illness, drug abuse, alcoholism, or drug addiction.
27. Pregnant or breastfeeding women.
28. Any past or current disease, treatment, or laboratory abnormality that may confound the study results, interfere with subject participation for the full duration of the study, or may not be in the best interest of the subject to participate in the study.
29. Local or systemic diseases caused by non-malignant tumors; or diseases or symptoms secondary to malignancy that may result in higher medical risk and/or uncertainty in survival assessment, such as tumor leukemic reaction (white blood cell count >20×109/L), cachexia (known weight loss exceeding 10% in the 3 months prior to screening), etc.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 2 years
  The proportion of patients whose tumor volume reduced by 30% and could maintain for more than 4 weeks, that is, the sum of the proportion of complete remission (CR) and partial remission (PR)

SECONDARY OUTCOMES:
Disease control rate （DCR) | 2 years
  The percentage of disease remission (including complete remission and partial remission, pr+cr) and stable disease (SD) in the number of evaluable cases after treatment
Duration of Response(DOR) | 2 years
  Remission duration refers to the time from the first CR or PR to disease progression.
Progression-Free-Survival （PFS） | 2 years
  Time from randomization to disease progression or death
Overall survival (OS) | 2 years
  The overall survival time of tumor patients
Adverse events | 2 years
  The incidence and severity of adverse events (AES) and clinically significant abnormal laboratory test results.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Shen, MD, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China